CLINICAL TRIAL: NCT04125511
Title: Characterizing IgG4-related Disease With 68Ga-FAPI PET/CT
Brief Title: Characterizing IgG4-RD With 68Ga-FAPI PET/CT
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PekingUMCHFAPI
Record Dates: First submitted 2019-08-28; First posted 2019-10-14 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: IgG4-related Disease
MeSH Terms: conditions — Immunoglobulin G4-Related Disease | interventions — 68Ga-FAPI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-FAPI, PET/CT (Experimental): Inject 68Ga-FAPI and then perform PET/CT scan.
  Interventions: Drug: 68Ga-FAPI

INTERVENTIONS:
Drug: 68Ga-FAPI — Intravenous injection of one dosage of 74-148 MBq (2-4 mCi) 68Ga-FAPI. Tracer doses of 68Ga-FAPI will be used to image lesions of IgG4-RD by PET/CT.
  Other Names: 68Ga-fibroblast activating protein inhibitors

SUMMARY:
68Ga-FAPI has been developed as a tumor-targeting agent as fibroblast activation protein is overexpressed in cancer-associated fibroblasts and some inflammation,such as IgG4-related disease.And it might be more sensitive than FDG in detecting a certain type of inflammations according to our preliminary research.Thus this prospective study is going to investigate whether 68Ga-FAPI PET/CT may be superior for diagnosis, therapy response assessment and follow-up of IgG4-related disease.

DETAILED DESCRIPTION:
Immunoglobulin G4-related disease (IgG4-RD) is an immune-mediated fibroinflammatory condition that is capable of affecting multiple organs. Common forms of presentation include:Type 1 (IgG4-related) autoimmune pancreatitis (AIP)，IgG4-related sclerosing cholangitis, major salivary gland enlargement or sclerosing sialadenitis; Orbital disease, often with proptosis and retroperitoneal fibrosis. The involved organs share a number of core pathologic features and striking clinical and serologic similarities, including tumor-like swelling of involved organs, a lymphoplasmacytic infiltrate enriched in IgG4-positive plasma cells, and a variable degree of fibrosis that has a characteristic "storiform" pattern. 68Ga-FAPI has been developed as a tumor-targeting agent as fibroblast activation protein is overexpressed in cancer-associated fibroblasts and it might be a pan-tumor PET agent. Recently we have reported a case of IgG4-related disease revealed by 68Ga-FAPI and 18F-FDG PET/CT which showed FAPI was not more tumor-specific than FDG, furthermore,it might be more sensitive than FDG in detecting a certain type of inflammations-like the pancreatic lesion. Thus this prospective study is going to investigate whether 68Ga-FAPI PET/CT may be superior for diagnosis, therapy response assessment and follow-up of IgG4-related disease.

ELIGIBILITY:
Inclusion Criteria:

* suspected or confirmed untreated IgG4-RD patients;
* 18F-FDG PET/CT within two weeks;
* signed written consent.

Exclusion Criteria:

* pregnancy;
* breastfeeding;
* known allergy against FAPI
* any medical condition that in the opinion of the investigator may significantly interfere with study compliance.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Metabolic parameters | through study completion, an average of 1 year
  Total Lesion Glycolysis (TLG) of focal lesions are measured on 68Ga-FAPI PET/CT.

SECONDARY OUTCOMES:
Diagnostic value | through study completion, an average of 1 year
  Diagnostic value of 68Ga-FAPI PET/CT for IgG4-RD in comparison with 18F-FDG PET/CT.
adverse events | through study completion, an average of 1 year
  Number of participants and kind of adverse events as a measure of safety.
Disease burden assessement | through study completion, an average of 1 year
  Correlation between disease burden assessed on 68Ga-FAPI PET/CT and clinical parameters for IgG4-RD.
FAPI expression and SUV | through study completion, an average of 1 year
  Correlation between FAPI expression and SUV in PET
Prediction value | through study completion, an average of 1 year
  Prediction value of 68Ga-FAPI PET/CT for IgG4-RD in therapy response assessment

CONTACTS AND LOCATIONS:
Overall Officials: Li Huo, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No